CLINICAL TRIAL: NCT00573820
Title: Phase 1 Study to Evaluate the Efficacy of Using Energy Specific Far Infrared Radiation Treatment for Prostate Cancer
Brief Title: Far Infrared Radiation Treatment for Prostate Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder & President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-PC-CTP1
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Prostatic Neoplasms
Keywords: Tumors or cancer of the prostate; Cancer of Prostate; Cancer of the Prostate; Neoplasms, Prostate; Neoplasms, Prostatic; Prostate Cancer; Prostate Neoplasms; Prostatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Radiation: Far Infrared Radiation

INTERVENTIONS:
Radiation: Far Infrared Radiation — Far Infrared Radiation (5μm to 20μm wavelength) for 30 to 40 minutes each treatment session.

SUMMARY:
A study to determine the use of far infrared radiation for the treatment of prostate cancer.

DETAILED DESCRIPTION:
Our initial assessment indicates that electromagnetic radiation of the central nervous system, the viscera and the endocrine system has the potential to cure a number of diseases, including prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Persons with Prostate, Bladder or Testicular Cancer.

Exclusion Criteria:

* None

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-01; Primary Completion 2008-02 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
The primary end point is to determine the therapeutic effects of far infrared radiation on Prostate Cancer. | 2 years and 6 months

SECONDARY OUTCOMES:
The secondary end point of the study is to evaluate the therapeutic effects of far infrared radiation on other types of cancer (Bladder and Testis). | 2 years and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.; Kwasi Donyina, Ph.D., Study Director — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada